CLINICAL TRIAL: NCT07404215
Title: Comparison of the Effects of Kinesio Taping and Dynamic Taping Applied to the Ankle on Vertical Jump, Balance, and Reaction Time in Basketball Players
Brief Title: Comparative Effects of Kinesio and Dynamic Taping on Ankle Performance in Basketball Players
Acronym: KT-DT-BB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Gamze Demircioğlu, Gamze Demircioglu, Atlas University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PI-DEMIRCIOGLU-2026
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Ankle Stability; Balance Performance; Vertical Jump Performance; Reaction Time; Basketball Players
Keywords: basketball; postural balance; ankle; reaction time; athletic tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping - Dorsiflexion Technique (Experimental): Participants assigned to this arm will receive ankle kinesio taping applied with the ankle positioned in dorsiflexion during tape application. The elastic tape will be applied from the plantar surface of the foot toward the calcaneus, Achilles tendon, and gastrocnemius muscle following standardized kinesio taping principles. This application technique aims to enhance proprioceptive input and neuromuscular control while allowing full ankle range of motion. Performance outcomes including balance, vertical jump, and reaction time will be assessed before and after the intervention.
  Interventions: Other: Kinesio Taping
- Kinesio Taping - Plantarflexion Technique (Experimental): Participants assigned to this arm will receive ankle kinesio taping applied with the ankle positioned in plantarflexion during tape application. The elastic tape will be applied using the same anatomical pathway and tension principles as the dorsiflexion technique, differing only in ankle positioning during application. This approach is intended to provide mechanical support and sensory feedback to the ankle joint without restricting movement. Balance, vertical jump performance, and reaction time will be evaluated before and after the intervention.
  Interventions: Other: Kinesio Taping

INTERVENTIONS:
Other: Kinesio Taping — Kinesio taping is an elastic therapeutic taping method applied to the ankle to support joint stability and neuromuscular control without restricting range of motion. In this study, kinesio taping is applied using two different application techniques that vary in ankle positioning during tape application.

SUMMARY:
This study aims to compare the effects of two different ankle taping methods-kinesio taping and dynamic taping-on balance, vertical jump performance, and reaction time in basketball players.

Basketball involves frequent jumping, rapid changes in direction, and single-leg balance, which place high demands on ankle stability. Reduced ankle stability may negatively affect athletic performance and increase the risk of injury. Taping methods are commonly used in sports practice to support the ankle joint and improve functional performance; however, limited evidence exists comparing different taping techniques in basketball players.

In this study, healthy male basketball players aged 18 to 30 years will receive both kinesio taping and dynamic taping applications in a crossover design, with a one-week interval between applications. Each participant will serve as their own control. Performance assessments will be conducted before and after each taping application.

Outcome measures include balance performance assessed using the Y-Balance Test, vertical jump performance assessed using a mobile application-based jump test, and lower extremity reaction time assessed using a visual-motor reaction task.

All procedures are non-invasive and associated with minimal risk. The findings of this study are expected to contribute to evidence-based taping strategies aimed at improving athletic performance and supporting ankle function in basketball players.

DETAILED DESCRIPTION:
This study is designed to compare the effects of kinesio taping and dynamic taping applied to the ankle joint on balance, vertical jump performance, and reaction time in basketball players.

Basketball is a high-intensity sport that involves frequent jumping, rapid acceleration and deceleration, sudden changes of direction, and single-leg balance tasks. During these activities, the ankle joint plays a critical role in load transmission, postural control, and neuromuscular coordination. Reduced ankle stability may negatively affect performance and increase the risk of injury in basketball players.

Taping techniques are commonly used in sports practice to support ankle stability, enhance proprioceptive input, and improve functional performance. Kinesio taping is proposed to facilitate neuromuscular control by increasing sensory feedback and modulating muscle activation, whereas dynamic taping is designed to absorb mechanical load, store elastic energy, and assist movement through elastic recoil. However, direct comparisons of these two taping methods in basketball players are limited.

This study uses a randomized, controlled, crossover design. Male basketball players aged 18 to 30 years who are actively competing at the professional level are planned to be included. All participants will provide written informed consent prior to participation. Each participant will receive both taping interventions, with a one-week washout period between applications, allowing each athlete to serve as their own control.

Kinesio taping and dynamic taping will be applied to the ankle and posterior lower leg according to standardized protocols described in the literature. All taping applications and performance assessments will be conducted by the same researcher, under standardized environmental conditions, and at similar times of day.

Outcome measures will be assessed immediately before and after each taping application to evaluate short-term effects. Vertical jump performance will be assessed using a validated mobile application, dynamic balance will be evaluated using the Y-Balance Test, and reaction time will be assessed using a visual-motor reaction time task focusing on lower extremity responses.

No invasive procedures will be performed during the study. All procedures are non-invasive and associated with minimal risk. The findings of this study are expected to contribute to evidence-based taping strategies aimed at improving athletic performance and supporting ankle function in basketball players.

ELIGIBILITY:
Inclusion Criteria:

* Male professional basketball players aged between 18 and 30 years
* Actively training and competing with a professional basketball team
* No history of lower extremity surgery within the past 6 months
* No acute lower extremity injury at the time of assessment
* Ability to perform single-leg jumping, balance, and reaction time tests
* Willingness to participate in the study and provide written informed consent

Exclusion Criteria:

* Presence of any acute musculoskeletal injury affecting the lower extremity
* History of ankle fracture, ligament rupture, or surgery within the past 6 months
* Neurological, vestibular, or systemic conditions affecting balance or motor performance
* Known allergy or skin reaction to adhesive taping materials
* Use of ankle bracing or taping within 48 hours prior to testing
* Inability to complete the assessment procedures

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Dynamic Balance Performance | Immediately before and immediately after each taping condition
  Dynamic balance performance will be assessed using the Y-Balance Test. Reach distances in the anterior, posteromedial, and posterolateral directions will be measured and normalized to limb length. A composite Y-Balance score will be calculated for each condition.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gencoglu C, Ulupinar S, Ozbay S, Turan M, Savas BC, Asan S, Ince I. Validity and reliability of "My Jump app" to assess vertical jump performance: a meta-analytic review. Sci Rep. 2023 Nov 17;13(1):20137. doi: 10.1038/s41598-023-46935-x. PMID 37978338
- [Result] Brinkman C, Baez SE, Quintana C, Andrews ML, Heebner NR, Hoch MC, Hoch JM. The Reliability of an Upper- and Lower-Extremity Visuomotor Reaction Time Task. J Sport Rehabil. 2020 Oct 7;30(5):828-831. doi: 10.1123/jsr.2020-0146. PMID 33027762
- [Result] Plisky P, Schwartkopf-Phifer K, Huebner B, Garner MB, Bullock G. Systematic Review and Meta-Analysis of the Y-Balance Test Lower Quarter: Reliability, Discriminant Validity, and Predictive Validity. Int J Sports Phys Ther. 2021 Oct 1;16(5):1190-1209. doi: 10.26603/001c.27634. eCollection 2021. PMID 34631241
- [Result] Powden CJ, Dodds TK, Gabriel EH. THE RELIABILITY OF THE STAR EXCURSION BALANCE TEST AND LOWER QUARTER Y-BALANCE TEST IN HEALTHY ADULTS: A SYSTEMATIC REVIEW. Int J Sports Phys Ther. 2019 Sep;14(5):683-694. PMID 31598406
- [Result] Nakajima MA, Baldridge C. The effect of kinesio(R) tape on vertical jump and dynamic postural control. Int J Sports Phys Ther. 2013 Aug;8(4):393-406. PMID 24175126
- [Result] Kodesh E, Benzoor MC, Dar G. Effect of dynamic tape on postural sway in individuals with chronic ankle instability. J Bodyw Mov Ther. 2021 Oct;28:62-67. doi: 10.1016/j.jbmt.2021.07.026. Epub 2021 Aug 8. PMID 34776201
- [Result] Biz C, Nicoletti P, Tomasin M, Bragazzi NL, Di Rubbo G, Ruggieri P. Is Kinesio Taping Effective for Sport Performance and Ankle Function of Athletes with Chronic Ankle Instability (CAI)? A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2022 Apr 29;58(5):620. doi: 10.3390/medicina58050620. PMID 35630037
- [Result] Alawna M, Mohamed AA. Short-term and long-term effects of ankle joint taping and bandaging on balance, proprioception and vertical jump among volleyball players with chronic ankle instability. Phys Ther Sport. 2020 Nov;46:145-154. doi: 10.1016/j.ptsp.2020.08.015. Epub 2020 Aug 29. PMID 32937273